CLINICAL TRIAL: NCT03733795
Title: Cerebral Perfusion During Intervention for Acute Respiratory Failure
Brief Title: Cerebral Perfusion and Acute Respiratory Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liverpool John Moores University (Other)
Collaborators: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 240082
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-10

CONDITIONS: Cerebral Blood Flow and Neonates During Acute Respiratory Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: 'Healthy babies' to establish 'normal' blood flow in neonates.
  Interventions: Other: TCD
- ECMO: Children undergoing extracorporeal membrane oxygenation for acute respiratory failure.
  Interventions: Other: TCD
- Conventional: Neonates undergoing conventional treatment for acute respiratory failure.
  Interventions: Other: TCD

INTERVENTIONS:
Other: TCD — Transcranial Doppler will be used to measure brain blood flow in the middle cerebral artery.

SUMMARY:
The most common reason for admitting babies and infants to an intensive care unit is due to respiratory distress (breathing difficulties). At present there are a number of different treatments for respiratory distress. These include drug treatments; non-invasive ventilation, where oxygen is given at high pressure to push it through the baby's lungs: ventilation where the baby is put on a breathing machine; or Extracorporeal Membrane Oxygenation (ECMO). This works by taking the blood from the body via a tube (usually) in the baby's neck, redirecting through a machine that oxygenates the blood, then returning it to the baby through another tube. Currently we know little about how different treatments have a different impact on brain perfusion (how much oxygen the brain gets). Using specialist, noninvasive ultrasound and doppler techniques, we are proposing to monitor the effect of these treatments on the brain.

DETAILED DESCRIPTION:
Following admission to Paediatric Intensive Care Unit, the clinical team will approach the parents of patients admitted with respiratory failure and introduce the research project. It is unlikely that parents will be have the capacity to provide meaningful full consent at this stage, as admission will be as an emergency. Therefore a two staged approach is proposed. Clinicians will act as gatekeepers to the parents. Parents/ patients deemed suitable for recruitment by clinicians will be provided with a brief explanation of the scan, and introduced to the researcher. Parents/patients may be deemed unsuitable should there be communication issues, legal issues (such as children in care) or clinical issues (where clinicians feel the patient is unlikely to survive and the research would be intrusive). With the parent's permission (documented in the research paperwork), scan data will collected from the patient. However, this will not be analysed or downloaded until after the second stage of consent. At a time deemed appropriate by the clinicians (based on clinical experience, this is expected to be within 24 hours of arrival) the researcher will provide a full explanation of the research and formally record parental consent on an approved form. At this point data generated will be downloaded and analysed. Should the parents refuse no more data will be collected. The measurements of brain blood flow will be taken using small probes located either side of the head. These will be held in place by either tape or a tubular bandage. Using an ultrasound images of the blood vessels (and flow) in the brain will also be measured at the same time. These measurements will be taken for 5-10 minutes on each occasion. Depending on treatment pathway, the data will be collected as follows: Measurements will be taken before treatment starts (in ECMO only). When the child is going onto treatment (during cannulation (ECMO) or intubation conventional)).

One hour after treatment has begun (ECMO only) 24 hours after treatment has started and then on a daily basis for the duration of treatment. During the weaning period where the patient is being prepared to come off treatment.

When the patient is being took off treatment (de-cannulation/extubation). One hour after they have been took off treatment. 24 hours after treatment has stopped. Not all the time points at which data will be collected will be applicable in every case.

Parents can withdraw consent at any point until data is analysed. No identifiable data will be recorded, apart from the consent forms.

ELIGIBILITY:
Inclusion Criteria:

* All neonates, infants and children undergoing treatment for acute respiratory failure.

Exclusion Criteria:

* Parents/guardians who do not wish for their child to participate.Parents/ guardians who are unable to provide written consent.
* Patients who clinicians feel are inappropriate to approach.

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: An estimation of 20, infants and children admitted with acute respiratory failure will be recruited from Alder Hey.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Differences in cerebral blood flow | 5 minutes for each scan
  Transcranial Doppler will be used to measure blood flow in the middle cerebral artery.

CONTACTS AND LOCATIONS:
Locations (1):
- Alder Hey Children's NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All information taken will be anonymised.